CLINICAL TRIAL: NCT02185859
Title: Effect of Perioperative Intravenous Lidocaine Infusion and Magnesium Infusion on the Functional Recovery After General Anesthesia in the Patients Undergoing Breast Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2014-0375
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Lidocaine; Magnesium; Mastectomy; Functional Recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Lidocaine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perioperative lidocaine infusion (Experimental)
  Interventions: Drug: Lidocaine
- Perioperative magnesium infusion (Experimental)
  Interventions: Drug: Magnesium Sulfate
- Noraml saline infusion (Active Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — The lidocaine group (Group L)- 1% lidocaine 40 mL is prepared in a 50 mL syringe; A bolus dose of the studied drugs are administered for 15 minutes immediately after a subject is brought into the operating room, and the vital signs are checked (from the beginning of anesthesia induction). Subsequently, an intravenous injection of the maintenance dose is continuously performed and later stopped just before transferring the subject to a recovery room. (Group L subjects are administered lidocaine 2 mg/kg for 15 minutes immediately after the anesthesia induction, and then lidocaine 2 mg/kg/h is continuously injected. The dose of lidocaine and magnesium in this study has been shown in previous studies to be safe and to have an analgesic effect.)
  Arms: Perioperative lidocaine infusion
Drug: Magnesium Sulfate — the magnesium group (Group M)- MgSO4 4g 40 mL is prepared in a 50 mL syringe.) A bolus dose of the studied drugs are administered for 15 minutes immediately after a subject is brought into the operating room, and the vital signs are checked (from the beginning of anesthesia induction). Subsequently, an intravenous injection of the maintenance dose is continuously performed and later stopped just before transferring the subject to a recovery room. The dose of magnesium in this study has been shown in previous studies to be safe and to have an analgesic effect.
  Arms: Perioperative magnesium infusion
Drug: Saline — the control group (Group C) - 0.9% normal saline 40 mL is prepared in a 50 cc syringe. A bolus dose of the studied drugs are administered for 15 minutes immediately after a subject is brought into the operating room, and the vital signs are checked (from the beginning of anesthesia induction). Subsequently, an intravenous injection of the maintenance dose is continuously performed and later stopped just before transferring the subject to a recovery room.Group C subjects are administered the same dose of normal saline.
  Arms: Noraml saline infusion

SUMMARY:
Postsurgical pain is a relevant side effect following surgery which increases the risk of various complications and delays postoperative patient recovery. Among the many types of surgeries, mastectomy causes not only acute but also chronic pain in many patients. Therefore, it is important to control pain and increase patients' recovery satisfaction following many kinds of operations by using as small an opioid analgesic dose as possible and adding a nonopioid analgesic to reduce the side effects of narcotic analgesics. Among nonopioid analgesics, lidocaine and magnesium are drawing attention, having been shown to be helpful in controlling postoperative pain by lowering pain hypersensitivity to surgical stimuli. An intraoperative intravenous injection of lidocaine has been reported to improve postoperative pain control by reducing postoperative pain and opioid consumption. Another report showed that an intraoperative intravenous injection of lidocaine improved the quality of postoperative functional recovery after general anesthesia in a laparoscopic cholecystectomy patient. In addition, a review article on the effect of intraoperative intravenous injection of magnesium found it to be an effective analgesic that may be added to conventional opioid-based therapy because it generally reduces opioid consumption, decreases pain assessment for 24 hours after surgery, and lacks severe side effects in relation to magnesium administration. However, there has been insufficient research comparing the intraoperative intravenous injection of lidocaine or magnesium in terms of which is more helpful for general functional recovery and decreased postoperative pain. Recently, the scope of research on anesthesia has come to embrace postanesthetic recovery; to help patients return to daily life, the research trend is now shifting from the improvement or resolution of a specific symptom to the measurement of general recovery. A widely used method to measure postoperative recovery is the Quality of Recovery 40 (QoR-40) survey.

Therefore, in this study, the researchers investigated the intraoperative intravenous injection of lidocaine and the intravenous injection of magnesium to compare these drugs' helpfulness in the functional recovery of mastectomy patients after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

-Patients aged between 20 and 65 who have undergone mastectomy due to breast cancer and of American Society of Anesthesiologists (ASA) Physical Status Class 1 or Class 2

Exclusion Criteria:

* Patients experiencing pain for any cause or taking an analgesic
* Pregnant patients
* Patients with severe heart, kidney, or liver disease
* Patients with a psychiatric or neurological disorder
* Patients with a contraindication or allergic response to lidocaine
* Patients with a contraindication or allergic response to magnesium

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The difference of QoR-40 global scores | 24 hours after mastectomy
  The investigators will evaluate the quality of recovery after general anesthesia by considering the global score (200 points in total) of QoR-40 surveys, which is obtained by summing the subtotal scores for emotional status, physical comfort, psychological support, physical independence, and pain. The QoR-40 administered 24 hours after the operation is the primary endpoint of this research.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, College of Medicine, Yonsei Health System, Yonsei Cancer Center, Seoul, Seoul, South Korea